CLINICAL TRIAL: NCT05046704
Title: Accuracy of Peripartum Ultrasound in the Prediction and Diagnosis of Obstetric Anal Sphincter Injuries
Brief Title: Peripartum Ultrasound in the Prediction and Diagnosis of OASIs
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Niven Abu Al-Foutouh Adly Shaban, Assistant Lecturer, Cairo University
Other Study IDs: peripartum US in OASIs.
Record Dates: First submitted 2021-09-13; First posted 2021-09-16 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Anal Sphincter Tear Complicating Delivery
Keywords: Obstetric Anal Sphincter Injuries; peripartum transperineal US; ano-vaginal distance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: peripartum transperineal Ultrasound — The anovaginal distance (AVD) will be measured by transperineal ultrasound ,The distance between the anal edge of the internal sphincter and the probe will then be measured in millimeters The ultrasound assessment of the anal sphincters at rest and during contraction will be performed postnatally using a dynamic 2-dimensional transperineal ultrasound with the patient in a supine position, an empty bladder.

SUMMARY:
To determine the value of peripartum scan measurement(s) in the prediction and diagnosis of Obstetric Anal Sphincter Injuries (OASIs)

DETAILED DESCRIPTION:
1.1.Obstetric Anal Sphincter Injuries (OASIs) Obstetric anal sphincter injuries (OASIs) are serious complications of vaginal birth with a reported incidence throughout Europe and globally, from 1-10% with recent UK data demonstrating a steadily rising incidence of this type of trauma over the past 12 years .

OASIs is one of the most significant risk factors for anal incontinence in young women as well as other complications of long-term dyspareunia and perineal pain.Despite optimal primary repair, approximately 39% of women who sustain an OASIs will suffer from anal incontinence. Several studies have reported a much higher risk of anal incontinence with subsequent deliveries and the potential for symptoms to progress with time.

1.2. Prediction of OASIs With the wealth of population based databases that are now available prediction models are being developed to assist in clinical decision making. Several large population based cohort studies have identified various independent risk factors for sustaining primary or recurrent OASIS. These include nulliparity, increased birth weight, operative vaginal delivery, persistent occipito-posterior position, prolonged pushing phase, induction of labour, use of epidural analgesia and shoulder dystocia, although findings across studies are contradictory.However there is paucity of information relating to the impact of risk factors that can only be known prior to the actual birth both on the likelihood of OASIs occurring de-novo and the usefulness of such information for counselling women at potential risk of sustaining a primary OASIs.

Although members of the investigators group have previously demonstrated that some of these prediction models have been suggested to have good discriminatory value, they do not necessarily confer a good clinical value. Although the model was useful in ruling out risk of OASIs in women with no risk factors, it was not as good in ruling-in an OASIS - that means that a women presenting with all of the known clinical risk factors cannot be differentiated at any higher risk than a women with a smaller subset of these risk factors. Hence limiting its clinical usability.

1.3. Ultrasound and OASIs management Transperineal and endoanal ultrasound scanning is currently used for the diagnosis and management of OASIs. Indeed, they form part of the recommended practice for determining the best mode of birth in pregnancies following OASIs.

Studies have also assessed some transperineal sonographic parameters, like the ano-vaginal distance (AVD), as a way of alerting clinicians to the possibility of OASIs. This measure has been used postnatally and a it was concluded that a short AVD could be a warning sign of possible external sphincter injury before suturing. The authors of this study suggested that an AVD of 20 mm seemed to indicate a cutoff level of the occurrence of external sphincter injury. Nevertheless, The authors of this study stressed on the need of further evaluation of their findings.

A However, to the investigators knowledge such parameter has not been assessed as an intrapartum tool, in combination with other radiological or clinical parameters, in the prediction of the risk of OASIs.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous .
2. Term, Vertex, Singleton living pregnancy.
3. Maternal age 18 years or over.
4. In labour.

Exclusion Criteria:

* Exclusion criteria are those who do not fit in the inclusion criteria.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Nulliparous, pregnant women in Term, Vertex, Singleton, 18 years or over, in labour.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Obstetric Anal Sphincter Injuries(OASIs) as diagnosed on clinical examination | baseline
  Detection the accuracy of peripartum transperineal US in prediction and diagnosis of obstetric anal sphincter injuries by measuring the ano vaginal distance in mm using vaginal probe of US and measuring the sub-pubic angle ueing 3D/4D probe of US intrapartum and using rolling technique postnatally for detection of occurrence of OASIs.

SECONDARY OUTCOMES:
1- Other degrees of perineal trauma | baseline
  to detect first and second degrees of perineal trauma by inspection and palpation to the perineal injuries.
2-Duration of second stage | baseline
  detection the time from fully dilated cervix to complete delivery of the fetus measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M Negm, Prof.Dr, Study Chair — Kasr Alainy Hospital-Cairo University.; Dalia S ZoElfakar, Assistant Prof.Dr, Study Chair — Kasr Alainy Hospital-Cairo University.; Mohamed F Youssef, : Lecturer Dr, Study Chair — Kasr Alainy Hospital-Cairo University.
Locations (1):
- Niven, Cairo, Egypt

REFERENCES:
- See also: Baghestan, E., Irgens, L.M., Børdahl, P.E., Rasmussen, S., (2010): Trends in Risk Factors for Obstetric Anal Sphincter Injuries in Norway. Obstet. Gynecol. 116, 25-34. — https://doi.org/10.1097/AOG.0b013e3181e2f50b
- See also: -Bellussi, F., Ghi, T., Youssef, A., Salsi, G., Giorgetta, F., Parma, D., Simonazzi, G., Pilu, G.,( 2017): The use of intrapartum ultrasound to diagnose malpositions and cephalic malpresentations. Am. J. Obstet. Gynecol. 217, 633-641. — https://doi.org/10.1016/j.ajog.2017.07.025
- See also: de Leeuw, J.., Struijk, P.., Vierhout, M.., Wallenburg, H.C.., (2001): Risk factors for third degree perineal ruptures during delivery. Br. J. Obstet. Gynaecol. 108, 383-387. https://doi.org/10.1016/S0306-5456(00)00090-5 — https://doi.org/10.1016/S0306-5456(00)00090-5
- See also: -Ismail, K.M.K.,( 2017): Perineal trauma at childbirth, Perineal Trauma at Childbirth. — http://doi.org/10.1007/978-3-319-14860-1